CLINICAL TRIAL: NCT00625846
Title: A Phase II Study of GW 786034 (Pazopanib) in Advanced Thyroid Cancer
Brief Title: Pazopanib Hydrochloride in Treating Patients With Advanced Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00198; NCI-2009-00198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC057H; CDR0000588044; 7627 (Other: Mayo Clinic); 7627 (Other: CTEP); N01CM00099 (NIH); N01CM62205 (NIH); P30CA015083 (NIH); NCT01648387 (obsolete NCT alias); NCT02653053 (obsolete NCT alias)
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Thyroid Gland Carcinoma; Stage III Differentiated Thyroid Gland Carcinoma AJCC v7; Stage III Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVA Differentiated Thyroid Gland Carcinoma AJCC v7; Stage IVA Thyroid Gland Anaplastic Carcinoma AJCC v7; Stage IVA Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVB Differentiated Thyroid Gland Carcinoma AJCC v7; Stage IVB Thyroid Gland Anaplastic Carcinoma AJCC v7; Stage IVB Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVC Differentiated Thyroid Gland Carcinoma AJCC v7; Stage IVC Thyroid Gland Anaplastic Carcinoma AJCC v7; Stage IVC Thyroid Gland Medullary Carcinoma AJCC v7; Thyroid Gland Anaplastic Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary; Thyroid Carcinoma, Anaplastic | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (DTC) (Experimental): Patients with differentiated thyroid cancer (DTC) receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride
- Cohort 2 (MTC) (Experimental): Patients with medullary thyroid cancer (MTC) receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pazopanib Hydrochloride
- Cohort 3 (ATC) (Experimental): Patients with anaplastic thyroid cancer (ATC) receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis
- Expansion Cohort (DTC) (Experimental): Patients with confirmed, differentiated thyroid cancer (DTC) who are thyroglobulin antibody negative receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Cohort 1 (DTC); Cohort 3 (ATC); Expansion Cohort (DTC)
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
  Arms: Cohort 1 (DTC); Cohort 2 (MTC); Expansion Cohort (DTC)

SUMMARY:
This phase II trial studies the side effects and how well pazopanib hydrochloride works in treating patients with advanced thyroid cancer. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety and efficacy of GW786034 (pazopanib hydrochloride) as a therapeutic in patients afflicted with differentiated, medullary and anaplastic thyroid cancers.

CORRELATIVE OBJECTIVES:

I. Assessment of the impact of therapy with GW786034 on serum/plasma vascular endothelial growth factor (VEGF) levels.

II. To explore the potential relationship between changes in thyroglobulin levels and tumor response in patients with advanced differentiated thyroid cancer known to be thyroglobulin antibody negative.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed differentiated, medullary or anaplastic thyroid cancer that is now advanced or metastatic; NOTE: patients with thyroid lymphomas or sarcomas are specifically excluded, as are patients with metastatic disease from other sites of origin to thyroid
* Patients with confirmed differentiated thyroid cancer to be enrolled in the expanded/additional differentiated thyroid cancer (DTC) cohort must be thyroglobulin antibody negative
* Zero, one or two prior therapeutic regimens (this includes cytotoxic plus non-cytotoxic therapeutic regimens)
* Absence of sensitivity to therapeutic radioiodine (differentiated only)
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan; NOTE: disease that is measurable by physical examination only is not eligible
* Life expectancy > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2 (Karnofsky >= 60%)
* Leukocytes > 3,000/mcL obtained =< 7 days prior to registration
* Absolute neutrophil count > 1,500/mcL obtained =< 7 days prior to registration
* Platelets > 100,000/mcL obtained =< 7 days prior to registration
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN) obtained =< 7 days prior to registration (if there is reason to believe that the patient has Gilbert's syndrome, the bilirubin can be fractionated; if the fractionated bilirubin is consistent with Gilbert's syndrome and there is no other possible explanation for the elevated indirect bilirubin, the patient may be eligible for the study if and only if the direct bilirubin is =< 1.5 X institutional ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 2.5 X institutional ULN obtained =< 7 days prior to registration
* Creatinine =< 1.5 X ULN obtained =< 7 days prior to registration
* Proteinuria =< + on urinalysis (may re-check) obtained =< 7 days prior to registration
* International normalized ratio (INR) =< 1.2 X the ULN obtained =< 7 days prior to registration
* Blood pressure (BP) < 140 mmHg (systolic) and < 90 mmHg (diastolic); initiation or adjustment of BP medication is permitted prior to registration provided that the average of three BP readings at a visit prior to registration is < 140/90 mmHg
* Objective evidence of tumor progression in the 6 month period prior to GW786034 initiation as assessed by:

  * Unequivocal progression of objectively measured disease on successive appropriate imaging (e.g. CT scan); in cases of uncertainty of tumor progression, the principal investigator of the study will be available to assist in decisions
* Women of child-bearing potential must have a negative serum pregnancy test =< 7 days prior to registration; NOTE: women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; effective contraception is required for all fertile participants in the trial
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to comply with the requirement of the study
* Willingness to donate blood for correlative marker studies; (only applicable to sites within the United States)

Exclusion Criteria:

* Anaplastic, differentiated, medullary: a total of > 2 prior therapeutic regimens (this total includes cytotoxic plus non-cytotoxic regimens); Note: enrollment of anaplastic, differentiated, and medullary patients who have had zero, one or two prior therapeutic regimens (cytotoxic plus non-cytotoxic regimens) is allowed - provided therapy ceased > 21 days prior to registration;

  * NOTE: the principal investigator of the study should be contacted in the event of uncertainty related patient eligibility based upon prior therapies
* Disease that is measurable by physical examination only
* Any of the following:

  * Radiotherapy =< 4 weeks prior to registration
  * Major surgery =< 4 weeks prior to registration
  * Radiotherapy to >= 25% of bone marrow
  * Concurrent therapy with octreotide unless tumor progression on this therapy has been demonstrated
* Any other ongoing investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW786034 (pazopanib) or other agents used in the study
* > +1 proteinuria (< 30 mg/dL) on two consecutive dipstick or other urine assessments taken at least 1 week apart; NOTE: (in cases where questions arise related to disparate proteinuria measurements, the study principal investigator [PI] should be consulted for assistance in determining patient study eligibility)
* Corrected QT interval (QTc) prolongation (defined as a QTc interval >= 480 msecs) or other significant electrocardiogram (ECG) abnormalities (e.g. frequent ventricular ectopy, evidence of ongoing myocardial ischemia); NOTE: the principal investigator of the study should be contacted in the event of uncertainty related patient eligibility based upon ECG changes
* Receiving cytochrome P450 (CYP) interactive concomitant medications; certain medications that act through the CYP450 system are specifically prohibited in patients receiving GW786034 (pazopanib) because in vitro data indicate that the agent has the potential to interact with the cytochrome P450 isoenzymes cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9) and cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); certain other agents should be used with caution
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain GSK786034 (pazopanib)
* Any of the following conditions:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, active diverticulitis, intra-abdominal abscess or gastrointestinal tract bleeding =< 28 days of registration
  * Any history of cerebrovascular accident (CVA) =< 6 months
  * Current use of therapeutic warfarin; Note: low molecular weight heparin and prophylactic low-dose warfarin (INR < 1.2 X ULN) are permitted; prothrombin time (PT)/partial thromboplastin time (PTT) must meet the inclusion criteria
  * History of myocardial infarction, cardiac arrhythmia, admission for unstable angina, cardiac angioplasty or stenting within the last 12 weeks
  * History of venous thrombosis in last 12 weeks
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; NOTE: a patient who has a history of class II heart failure and is asymptomatic on treatment may be considered eligible
  * History of bleeding disorder, including patients afflicted with hemophilia, disseminated intravascular coagulation, or any other abnormality of coagulation potentially predisposing patients to bleeding
  * Poorly controlled depression or anxiety disorder, or recent (=< 6 months) suicidal ideation
* Known active and/or untreated brain metastases and/or brain metastases requiring ongoing therapy (e.g. corticosteroids); NOTE: (because of the poor prognosis often associated with brain metastases and because of the potential risk of bleeding in active brain metastases associated with multi-targeted tyrosine kinase inhibitor therapy, patients with active and/or untreated brain metastases and/or those with brain metastases requiring ongoing therapy - e.g. corticosteroids - are excluded from trial enrollment; enrollment will, however, be permitted in cases of patients with longstanding treated and inactive brain metastases not requiring ongoing therapy, providing that stability of brain metastases has been demonstrated for a period of 3 months or greater as assessed by intracranial imaging - and providing that there is no indication of increased vascularity of the treated metastases by magnetic resonance imaging (MRI) imaging conducted =< 14 days prior to registration; when questions arise related to these criteria, the PI of the trial, Dr. Keith Bible, should be contacted for assistance on eligibility)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would or might reasonably be expected to limit compliance with study requirements
* Pregnant women; NOTE: (breastfeeding should be discontinued if the mother is treated with GW786034/pazopanib)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy; NOTE: (appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated)
* Receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of GW786034 (pazopanib); NOTE: the eligibility of patients will be determined following review of their case by the principal investigator; efforts should be made to switch patients who are taking enzyme-inducing anticonvulsant agents to other medications
* Receiving any concomitant medications that are associated with a risk of QTc prolongation and/or Torsades de Pointes; NOTE: these medications should be discontinued or replaced with drugs that do not carry these risks, if possible

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-02-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith C Bible, Principal Investigator — Mayo Clinic
Locations (22):
- United States (16):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China
- Singapore (3):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre, Singapore
  - Johns Hopkins Singapore, Singapore
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Bible KC, Menefee ME, Lin CJ, Millward MJ, Maples WJ, Goh BC, Karlin NJ, Kane MA, Adkins DR, Molina JR, Donehower RC, Lim WT, Flynn PJ, Richardson RL, Traynor AM, Rubin J, LoRusso PM, Smallridge RC, Burton JK, Suman VJ, Kumar A, Voss JS, Rumilla KM, Kipp BR, Chintakuntlawar AV, Harris P, Erlichman C. An International Phase 2 Study of Pazopanib in Progressive and Metastatic Thyroglobulin Antibody Negative Radioactive Iodine Refractory Differentiated Thyroid Cancer. Thyroid. 2020 Sep;30(9):1254-1262. doi: 10.1089/thy.2019.0269. Epub 2020 Jul 29. PMID 32538690
- [Derived] Bible KC, Suman VJ, Molina JR, Smallridge RC, Maples WJ, Menefee ME, Rubin J, Sideras K, Morris JC 3rd, McIver B, Burton JK, Webster KP, Bieber C, Traynor AM, Flynn PJ, Goh BC, Tang H, Ivy SP, Erlichman C; Endocrine Malignancies Disease Oriented Group; Mayo Clinic Cancer Center; Mayo Phase 2 Consortium. Efficacy of pazopanib in progressive, radioiodine-refractory, metastatic differentiated thyroid cancers: results of a phase 2 consortium study. Lancet Oncol. 2010 Oct;11(10):962-72. doi: 10.1016/S1470-2045(10)70203-5. Epub 2010 Sep 17. PMID 20851682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
Started | 39 | 35 | 16 | 62
Completed | 37 | 35 | 15 | 60
Not Completed | 2 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All patients that registered and evaluable for any of the endpoints were included in this summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC) | Total
Number analyzed (Participants) | 37 | 35 | 15 | 60 | 147
Age, Continuous [Median (Full Range); unit: years] | 63 [23 to 79] | 60 [48 to 70] | 66 [45 to 77] | 60 [51 to 69] | 61 [23 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 10 | 27 | 62
  Male | 19 | 28 | 5 | 33 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3 | 6
  Not Hispanic or Latino | 29 | 33 | 12 | 57 | 131
  Unknown or Not Reported | 7 | 1 | 2 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 2 | 17 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 4 | 4
  White | 35 | 28 | 12 | 37 | 112
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Singapore | 1 | 3 | 2 | 3 | 9
  United States | 35 | 26 | 13 | 38 | 112
  China | 0 | 1 | 0 | 0 | 1
  Taiwan | 0 | 3 | 0 | 10 | 13
  Australia | 1 | 2 | 0 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (in Cohorts 1-3)
Description: The tumor response rate is defined as the percentage of eligible patients who fulfill RECIST 1.0 for a complete or partial response at two consecutive assessments at least 8 weeks apart for patients in Cohorts 1-3. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Population: All patients in Cohort 1, Cohort 2, and Cohort 3 that received treatment and were eligible for response assessment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1 (DTC): Patients with differentiated thyroid cancer (DTC) receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.> > Laboratory Biomarker Analysis: Correlative studies>
  > Pazopanib Hydrochloride: Given PO
- Cohort 2 (MTC): Patients with medullary thyroid cancer (MTC) receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Pazopanib Hydrochloride: Given PO
- Cohort 3 (ATC): Patients with anaplastic thyroid cancer (ATC) receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Laboratory Biomarker Analysis: Correlative studies
- Expansion Cohort (DTC): Patients with confirmed, differentiated thyroid cancer (DTC) who are thyroglobulin antibody negative receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.> > Laboratory Biomarker Analysis: Correlative studies>
  > Pazopanib Hydrochloride: Given PO
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
Number analyzed (Participants) | 37 | 35 | 15 | 0
percentage of participants | 49 [35 to 68] | 14 [6 to 28] | 0 [0 to 22] |

2. Primary Outcome: Confirmed Tumor Response (in the Differentiated Thyroid Cancer Expansion Cohort)
Description: The confirmed tumor response rate is defined as the percentage of eligible patients who fulfill RECIST 1.0 for a complete or partial response at two consecutive assessments at least 8 weeks apart for patients with differentiated thyroid cancer who are thyroglobulin antibody negative. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Population: All patients that registered to the Differential Thyroid Expansion cohort and were evaluable for response assessment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
Number analyzed (Participants) | 0 | 0 | 0 | 60
percentage of participants |  |  |  | 37 [25 to 50]

3. Secondary Outcome: Toxicity as Measured by the Percentage of Patients Reporting a Grade 3+ Adverse Event Deemed Possibly, Probably, or Definitely Related to Treatment
Description: Toxicity (defined as grade 3+ adverse events deemed possibly, probably, or definitely related to treatment) will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0. The percentage of patients with grade 3+ adverse events deemed possibly, probably, or definitely related to treatment are reported for patients in Cohorts 1-3.
Time Frame: Up to 3 years
Population: All patients that received protocol treatment and were assessed for adverse events are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
Number analyzed (Participants) | 38 | 35 | 15 | 61
percentage of participants | 40 | 46 | 53 | 53

4. Secondary Outcome: Progression-Free Survival at 6 Months (Cohorts 1 and 2 Only)
Description: Progression free survival at 6 months (PFS6) is defined as the proportion of patients alive and without progression at 6 months. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0.
Time Frame: Time from registration to the date of progression or last follow-up, whichever comes first, assessed up to 6 months
Population: All patients in Cohort 1 and Cohort 2 that received treatment and were eligible for response assessment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
Number analyzed (Participants) | 37 | 35 | 0 | 0
proportion of participants | .71 [.58 to .87] | .686 [.548 to .858] |  |

5. Secondary Outcome: Progression-Free Survival at 3 Months (Cohort 3 Only)
Description: Progression free survival at 3 months (PFS6) is defined as the proportion of patients alive and without progression at 3 months. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0.
Time Frame: Time from registration to the date of progression or last follow-up, whichever comes first, assessed up to 3 months
Population: All patients from Cohort 3 that were treated and evaluable for response were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
Number analyzed (Participants) | 0 | 0 | 15 | 0
proportion of participants |  |  | .267 [.115 to .617] |

6. Other Pre Specified Outcome: Change in Blood Markers for Angiogenesis
Description: Blood markers for angiogenesis including levels of free VEGF, free GW786034, and GW786034/VEGF complexes will be evaluated before and during therapy. Changes in these levels will largely be explored in a graphical manner as well as exploring any potential relationships between these levels and clinical outcome such as response or progression-free rate and toxicity incidence.
Time Frame: Baseline to up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Proportion of Patients With Differentiated Thyroid Cancer and Medullary Thyroid Cancer Who Have Not Failed Treatment at 6 Months (3 Months for Anaplastic Thyroid Cancer)
Description: The proportion of patients who have not failed treatment due to disease progression, adverse reactions, refusal for further participation, or who went on to alternate therapy at 6 months (3 months for anaplastic thyroid cancer patients) will be calculated and summarized independently within each of the patient groups. Assuming that the incidence of response is binomially distributed, 90% binomial confidence intervals will also be calculated.
Time Frame: Up to 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause. The median is estimated using the Kaplan-Meier estimator.> Estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to date of last follow-up or death due to any cause, assessed up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Time to Treatment Failure
Description: Estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the date the patient discontinues treatment, assessed up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Time to Subsequent Therapy
Description: Estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression (PD) is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by >= 50% of previously involved sites from nadir). Duration of response will be assessed.
Time Frame: Time from registration to the date the patient discontinues treatment, assessed up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of every 28 day cycle, up to 84 cycles.
Description: Adverse events were collected at the end of every 28 day cycle, up to 84 cycles.
Arm/Group | Cohort 1 (DTC) | Cohort 2 (MTC) | Cohort 3 (ATC) | Expansion Cohort (DTC)
All-Cause Mortality (participants affected / at risk) | 3/38 | 0/35 | 1/15 | 4/61
Serious Adverse Events (participants affected / at risk) | 21/38 | 18/35 | 9/15 | 31/61
Other Adverse Events (participants affected / at risk) | 38/38 | 35/35 | 15/15 | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (DTC) (N=38) | Cohort 2 (MTC) (N=35) | Cohort 3 (ATC) (N=15) | Expansion Cohort (DTC) (N=61)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (20) | 1 (1) | 0 (0) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0) | 4 (6)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Wound infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bilirubin increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (5) | 0 (0) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (1) | 2 (4) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 9 (11) | 4 (6) | 0 (0) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (10) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (6) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (21) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (17) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 5 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (15) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (20) | 2 (3) | 0 (0) | 2 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (21) | 0 (0) | 0 (0) | 6 (8)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (DTC) (N=38) | Cohort 2 (MTC) (N=35) | Cohort 3 (ATC) (N=15) | Expansion Cohort (DTC) (N=61)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (70) | 14 (103) | 7 (11) | 33 (182)
Palpitations (Cardiac disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (13)
Conjunctival disorder (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 4 (12)
Constipation (Gastrointestinal disorders) | 3 (6) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 28 (294) | 29 (380) | 7 (17) | 48 (505)
Dry mouth (Gastrointestinal disorders) | 2 (8) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (5) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (6) | 0 (0) | 1 (2)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 29 (166) | 19 (94) | 6 (11) | 28 (136)
Oral hemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (4) | 1 (6) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 18 (41) | 9 (31) | 3 (3) | 20 (71)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 35 (275) | 29 (286) | 12 (28) | 50 (479)
Fever (General disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 14 (72) | 4 (16) | 1 (2) | 12 (21)
Alkaline phosphatase increased (Investigations) | 6 (8) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 16 (72) | 15 (72) | 6 (10) | 30 (97)
Bilirubin increased (Investigations) | 8 (20) | 3 (13) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (17) | 0 (0) | 0 (0) | 2 (2)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 16 (51) | 14 (60) | 4 (11) | 33 (221)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (21) | 1 (6) | 6 (19)
Neutrophil count decreased (Investigations) | 14 (26) | 8 (27) | 1 (2) | 28 (142)
Platelet count decreased (Investigations) | 14 (41) | 10 (38) | 1 (1) | 19 (68)
Serum cholesterol increased (Investigations) | 2 (2) | 3 (6) | 0 (0) | 1 (1)
Weight loss (Investigations) | 12 (75) | 5 (9) | 0 (0) | 6 (44)
Anorexia (Metabolism and nutrition disorders) | 23 (93) | 20 (91) | 8 (14) | 28 (133)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (18) | 3 (8) | 0 (0) | 1 (2)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 5 (21) | 2 (5) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 2 (3) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (10) | 1 (1) | 2 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (11) | 3 (7) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 2 (2) | 0 (0) | 4 (6)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Olfactory nerve disorder (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (31) | 8 (42) | 0 (0) | 12 (40)
Taste alteration (Nervous system disorders) | 22 (128) | 5 (19) | 2 (2) | 9 (33)
Agitation (Psychiatric disorders) | 0 (0) | 4 (9) | 1 (2) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 7 (26) | 1 (1) | 7 (25)
Depression (Psychiatric disorders) | 2 (3) | 5 (31) | 0 (0) | 8 (28)
Euphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 4 (9) | 2 (4) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 10 (79) | 15 (27) | 8 (10) | 27 (121)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 0 (0) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (11) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (14) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (79) | 2 (8) | 0 (0) | 3 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (7) | 0 (0) | 0 (0)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (6) | 0 (0) | 8 (10)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (7) | 1 (8) | 0 (0) | 1 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (9) | 1 (4) | 0 (0) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 28 (337) | 22 (339) | 5 (10) | 42 (490)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hot flashes (Vascular disorders) | 2 (14) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 21 (81) | 20 (239) | 8 (10) | 46 (497)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT00625846/Prot_SAP_000.pdf